CLINICAL TRIAL: NCT02099383
Title: A Phase III Trial of BUN/Cr-based Hydration Therapy to Reduce Stroke-in-evolution and Improve Short-term Functional Outcomes for Dehydrated Patients With Acute Ischemic Stroke
Brief Title: BUN/Cr-based Hydration Therapy to Improve Outcomes for Dehydrated Patients With Acute Ischemic Stroke.
Acronym: HYDO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPRPG6D0011
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2018-11

CONDITIONS: Stroke; Dehydration
Keywords: Stroke; Dehydration; Fluid Therapy
MeSH Terms: conditions — Stroke; Dehydration | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal saline, bolus (Active Comparator): Patients of study group will receive intravenous normal saline 20cc per kilogram of body weight, one third of which will be given as a bolus followed by delivery of the remaining two third as a constant infusion over a period of 8 hours.
  Interventions: Other: normal saline
- normal saline, control (No Intervention): Patients of control group will receive intravenous normal saline 60 cc per hour.

INTERVENTIONS:
Other: normal saline — intravenous normal saline 20cc per kilogram of body weight over a period of 8 hours
  Arms: normal saline, bolus

SUMMARY:
The investigators' preliminary findings suggest that providing patients with acute ischemic stroke hydration therapy on the basis of their presenting BUN/Cr ratio may help reduce the occurrence of stroke-in-evolution(SIE) and therefore improve prognosis.

The trial will be carried out in two parts. Part 1 assesses the rate of stroke-in-evolution 72 hours after the onset of stroke as a measure of the activity of BUN/Cr ratio based hydration therapy. Part 2, The investigators use two outcome measures, including Barthel index, and modified Rankin scale for neurological evaluation to assess whether BUN/Cr ratio based hydration therapy results in sustained clinical benefit at three months.

DETAILED DESCRIPTION:
The investigators have recently reported a novel finding that the blood urea nitrogen (BUN)/creatinine (Cr) ratio, a marker of hydration status, was an independent predictor of SIE among patients who had suffered acute ischemic stroke. The investigators found that patients who had a BUN/Cr ratio ≥ 15 were 3.4-fold more likely to experience SIE than patients who had a BUN/Cr ratio < 15. The ratio of SIE was 13.9% in all patients, with 20% in patients who had a BUN/Cr ratio ≥ 15 and 8.3% in patients who had a BUN/Cr ratio < 15. Among the patients presenting with acute ischemic stroke, 37% of them had a BUN/Cr ratio ≥ 15.

The investigators' recent pilot study was designed to determine if providing hydration therapy, specifically intravenous saline infusion, to patients with a blood urea nitrogen/creatinine ratio (BUN/Cr) ≥15 reduces the occurrence of SIE after acute ischemic stroke. Patients in the hydration group received a significantly larger (all P < 0.001) median volume of infused saline than patients in the control group. And this allowed 82% of the patients to maintain their BUN/Cr ratio <15 in first 8 hours. The proportion of patients who experienced SIE was significantly lower in the hydration group compared with the control group.

Dehydration, as indicated by an increased BUN/Cr ratio, is known to be relatively common among patients who have experienced stroke. According to the result of our pilot study, a hydration strategy with intravenous 20 cc per kilogram of body weight normal saline in first 8 hours was safe and effective to prevent dehydration related early neurological deterioration.

In this study, the investigators conduct a randomized double-blind control trial to test the hypothesis that whether BUN/Cr ratio based hydration therapy has clinical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke diagnosed by the clinical presentations and brain imaging is confirmed by a stroke care specialist.
2. has a measurable neurologic deficit according to the National Institutes of Health Stroke Scale (NIHSS)
3. the time between the onset of neurological symptoms and starting therapy are less than 12 hours
4. admission BUN/Cr≧15

Exclusion Criteria:

1. no informed consent obtained
2. initial NIHSS >15
3. prepared for or received fibrinolytic therapy
4. prepared for or received surgical intervention with 14 days
5. congestive heart failure according to past history or Framingham criteria
6. history of liver cirrhosis or severe liver dysfunction (alanine aminotransferase or aspartate aminotransferase > x 3 upper normal limit)
7. admission blood Cr >2 mg/dl
8. initial systolic blood pressure <90 mmHg
9. fever with core temperature >=38°C
10. indication of diuretics for fluid overload
11. any conditions needed more aggressive hydration or blood transfusion
12. cancer under treatment
13. life expectancy or any reasons for follow-up < 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2014-04; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
rate of stroke-in-evolution | 72 hours
  Stroke-in-evolution is defined as a deterioration from base line in the score on the NIHSS by 4 or more points.

SECONDARY OUTCOMES:
rate of favorable outcome | three months
  Scores of >=60 on the Barthel index, <=2 on the modified Rankin scale are considered to indicate a favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Leng C Lin, MD, Principal Investigator — Department of Emergency Medicine, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin LC, Yang JT, Weng HH, Hsiao CT, Lai SL, Fann WC. Predictors of early clinical deterioration after acute ischemic stroke. Am J Emerg Med. 2011 Jul;29(6):577-81. doi: 10.1016/j.ajem.2009.12.019. Epub 2010 Apr 2. PMID 20825831
- [Derived] Lin LC, Lee TH, Huang YC, Tsai YH, Yang JT, Yang LY, Pan YB, Lee M, Chen KF, Hung YC, Cheng HH, Lee IN, Lee MH, Chiu T, Chang YJ, Goh ZNL, Seak CJ. Enhanced versus standard hydration in acute ischemic stroke: REVIVE-A randomized clinical trial. Int J Stroke. 2024 Oct;19(9):1010-1019. doi: 10.1177/17474930241259940. Epub 2024 Jul 31. PMID 38785314